CLINICAL TRIAL: NCT02024737
Title: A Pilot Study to Establish the Sensitivity of MR Imaging Markers to Changes in Regional Lung Function and Gas Washout in Patients With Mild-moderate COPD
Brief Title: SILO2 (Signal Intensity Lung washOut)
Acronym: SILO2
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: STH17337
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Moderate-Severe COPD: Patients with moderate to severe COPD, as defined by GOLD 2-3 (The GOLD classifications are the main method doctors use to describe the severity of COPD.
  GOLD is short for the Global Initiative for Chronic Obstructive Lung Disease, a collaboration between the National Institutes of Health and the World Health Organization)
  Interventions: Other: MRI lung imaging (not an intervention per se but the focus of the study)

INTERVENTIONS:
Other: MRI lung imaging (not an intervention per se but the focus of the study) — The purpose of this pilot study is to determine short and long term reproducibility of a comprehensive set of functional imaging data; using hyperpolarised gas MRI, conventional MRI and lung physiology measurements in patients with moderate to severe COPD. In addition,how sensitive the imaging techniques are to changes in lung function after treatment with a standard (bronchodilator) inhaler will also be assessed (the bronchodilator foradil is a non-investigative medicinal product as it is a medicine with a known effect which will be used to induce a known response).
  This pilot study will serve as a platform for future larger scale studies, aimed at better understanding of and intervention in early COPD.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a leading and still increasing cause of disease and death worldwide, affecting those in both developed and developing countries. This imparts a massive burden of ill health, in turn imposing huge healthcare costs to society.

For effective treatment of COPD (as opposed to providing short term relief) early disease must be targeted. The small airways of the lung (those less than 2mm) are the first affected in COPD, but current methods to assess their function are relatively insensitive. There is therefore a need for new, accurate methods for detection of small airway dysfunction with sensitivity to shortterm change and regional discrimination.

In previous studies with hyperpolarised (HP) 3He MRI in smokers with normal pirometry and patients with early stage COPD, we showed sensitivity to early changes in lung ventilation and structure. The hyperpolarised gas MRI technique is safe. In particular, the lack of ionizing radiation permits patients to be imaged on multiple occasions. This and its inherent sensitivity to regional lung ventilation and function make it an ideal imaging tool for the assessment of novel lung therapies for diseases of the small airways.

The purpose of this pilot study is to determine short and long term reproducibility of a comprehensive set of functional imaging data; using hyperpolarised gas MRI, conventional MRI and lung physiology measurements in patients with moderate to severe COPD.

In addition,how sensitive the imaging techniques are to changes in lung function after treatment with a standard (bronchodilator) inhaler will also be assessed.

This pilot study will serve as a platform for future larger scale studies, aimed at better understanding of and intervention in early COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥40 years, who have signed an Informed Consent Form prior to initiation of study related procedures.
* Current or exsmokers who have a smoking history of at least 10 pack years. (Ten pack years are defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years etc.)
* Clinical diagnosis of COPD with a post bronchodilator FEV1 30-80% of personal predicted, according to GOLD (Global Initiative for Chronic Obstructive Lung Disease) guidelines.

Exclusion Criteria:

* Patients with a contra-indication to MRI scanning: i.e. patients who are non MRI compatible (ferro-magnetic metallic implants, pacemakers) as per the MRI questionnaire used in clinical practice by the Unit of Academic Radiology, Royal Hallamshire Hospital, or who are unable to tolerate the MRI.
* Patients with renal conditions (as described in the Gd-DTPA (Gadovist) Summary of Product Characteristics) in which administration of Gd-DTPA MR vascular contrast agent would pose a risk.
* Patients contraindicated for treatment with, or having a history of reactions/ hypersensitivity to any of the following inhaled drugs, drugs of a similar class or any component thereof:

  * long and short acting beta-2 agonists
  * sympathomimetic amines
  * lactose or any of the other excipients
* Resting oxygen saturation of <90% on air as determined by pulse oximetry.
* Women of child bearing potential, not using effective methods of contraception.
* Pregnant women or nursing mothers (pregnancy confirmed by positive urine pregnancy test).
* Inability to understand or comply with study procedures; including patients unable to use a dry powder inhaler (e.g. single dose dry powder inhaler Aerolyzer®) device.
* Significant pulmonary pathology other than COPD.
* Previous lung surgery.
* Patients taking oral theophyllines, PDE4 inhibitors or leukotriene antagonists, or on maintenance treatment with oral steroids.
* Patients who are participating in the active phase of a supervised pulmonary rehabilitation program.
* Patients with a history of long QT syndrome or whose QTc measured (Fridericia method) is prolonged (>450 ms for males and females) or a history of dysrhythmia other than established chronic atrial fibrillation.
* Subjects with unstable cardiac disease which in the opinion of the investigator exposes them to significant additional risk. .
* Heart failure which is either unstable or the predominant cause of the subject's dyspnea.
* Patients who, in the judgment of the investigator, had a clinically relevant laboratory abnormality or a clinically significant condition such as (but not limited to):

  * Any condition which might compromise patient safety or compliance, interfere with evaluation, or preclude completion of the study.
  * Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of study enrollment (whichever is longer).
  * Patients unable to use a dry powder inhaler (e.g. single dose dry powder inhaler Aerolyzer®) device.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from COPD clinics in Sheffield, the surrounding area and the nurse-led clinics running alongside them, by open advertisement, after pulmonary rehabilitation, and via invitation by their local GP. The target is to recruit 6 subjects within 4 months.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Reproducibilityof 3He and 129Xe MRI lung ventilation imaging as measured by Bland-Altman statistical analysis of reproducibility | 48 hours
  Measure of short-term reproducibility of MRI imaging
Reproducibilityof 3He and 129Xe MRI lung ventilation imaging as measured by Bland-Altman statistical analysis of reproducibility | 21 days
  Measure of long-term reproducibility of MRI imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom